CLINICAL TRIAL: NCT05336526
Title: Evaluation of the Safety and Performance of SYMATESE AESTHETICS ESTYME® MATRIX Round Microtextured Silicone Gel-Filled Breast Implants in the Breast Augmentation, Primary Intention (EMMA Study)
Brief Title: Evaluation of the Safety and Performance of SYMATESE AESTHETICS ESTYME® MATRIX Round Microtextured Silicone Gel-Filled Breast Implants in the Breast Augmentation
Acronym: EMMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Symatese Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLIN PMI-004
Record Dates: First submitted 2022-03-23; First posted 2022-04-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Bilateral Breast Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESTYME® MATRIX Round Microtextured Silicone Gel-Filled Breast Implants (Experimental): Participants who meet the requirements for bilateral breast augmentation in primary intention and have been implanted with ESTYME® MATRIX Round Microtextured Silicone Gel-Filled Breast Implants
  Interventions: Device: ESTYME® MATRIX Round Microtextured Silicone Gel-Filled Breast Implants

INTERVENTIONS:
Device: ESTYME® MATRIX Round Microtextured Silicone Gel-Filled Breast Implants — Bilateral brest augmentation in primary intention

SUMMARY:
The purpose of this study is to collect clinical data to evaluate the safety and performance of ESTYME® MATRIX Round microtextured breast implants in patients who receive these silicone gel-filled implants as part of their breast augmentation surgery in primary intention. This study also aims to measure patient and surgeon satisfaction.

An initial study of all ESTYME® MATRIX implants was conducted between 2018 and 2021. The purpose of the current EMMA study is to complete the data from this first study on a larger number of implants, and only on the ESTYME® MATRIX Round Microtextured Silicone Gel-Filled Breast Implants range for primary intention breast augmentation, with a view to obtaining marketing authorization (CE marking).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years
2. Eligible for bilateral breast augmentation in primary intention

   1. general breast enlargement for cosmetic purposes
   2. surgical correction of various congenital or acquired anomalies such as amastia, aplasia, hypomastia, hypoplasia, asymmetries*, Poland's syndrome*, ptosis … * correction of asymmetries and Poland's Syndrome with concomitant augmentation of the second breast (bilateral implantation)
3. Signature of Patient Information Consent (PIC) & willingness to comply with the protocol assessments and follow up visits
4. Affiliation to the social security regime

Exclusion Criteria:

1. Local or systemic infection or abscess anywhere in the body
2. Existing carcinoma or pre-carcinoma of the breast with or without treatment
3. History of subcutaneous mastectomy
4. Subject with previous tissue expansion
5. Diagnosis of active cancer of any type
6. Pregnant subject or intending to become pregnant within three (3) months after the implant procedure (women of childbearing potential must use effective contraception from 1 month before the implantation procedure until 3 months after the implantation procedure)
7. Has breastfed within three (3) months the implant surgery, or is still breastfeeding
8. Tissue characteristics determined as clinically inadequate or unsuitable by the surgeon (i.e. tissue damage resulting from radiation, inadequate tissue or compromised vascularity, known wound healing complications)
9. Has been previously implanted with a silicone implant or history of failure following cosmetic augmentation
10. History of autoimmune disease such as, but not limited to, lupus and scleroderma
11. Any condition or treatment for any condition which, in the opinion of the investigator, may constitute an unwarranted surgical risk (e.g. severe lung or cardiac disease, unstable medical conditions, anaesthesia allergy, heavy smokers…)
12. Anatomic or physiologic abnormality which could result to significant post-operative complications
13. History of sensitivity to foreign materials or known allergy to any component of the ESTYME® MATRIX Round Microtextured Silicone Gel-Filled Breast Implant
14. Known alcohol abuse or history of alcohol abuse
15. Psychological instability
16. Underlying disease (HIV-positive, heart failure, renal insufficiency, diabetes, hypertension)
17. Implanted metal or metal devices, history of claustrophobia, or other condition that would make a magnetic resonance imaging (MRI) scan prohibitive
18. Unwilling to undergo any further surgery for revision
19. Unrealistic/unreasonable expectations that entail a risk for the surgical procedure
20. Participating in another clinical study or within exclusion period of a previous clinical study as determined by the investigator
21. Has sociological, cultural or geographical factors which could interfere with evaluation or completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety : Incidence of implant and/or procedure-related adverse events/complications | 3 months post-procedure
  Safety endpoint will be assessed by the incidence of implant and/or procedure-related adverse events/complications at 3 months post implant

SECONDARY OUTCOMES:
Safety : Incidence of all AEs/SAEs | 1 year post-procedure
  Safety endpoint will be assessed by the incidence of all AEs/SAEs at 1 year post-procedure
Safety : Incidence of all AEs/SAEs | 2 years post-procedure
  Safety endpoint will be assessed by the incidence of all AEs/SAEs at 2 years post-procedure
Performance, Implant procedure Success: Surgeon comfort evaluation with procedure duration | at the implant procedure
  Evaluation of surgeon 's satisfaction with procedure duration (5 options: Definitely satisfied, Satisfied, Somewhat satisfied, Somewhat dissatisfied, Definitely dissatisfied)
Performance, Implant procedure Success: Surgeon comfort evaluation with size incision | at the implant procedure
  Evaluation of surgeon 's satisfaction with size of incision (5 options: Definitely satisfied, Satisfied, Somewhat satisfied, Somewhat dissatisfied, Definitely dissatisfied)
Performance, Implant procedure Success: Assessment of implant placement and deformation | 3 months post-procedure
  Assessment of the implant correct placement (absence of visible deformation of the gel) at 3 months
Performance :Surgeon comfort evaluation with comfort level for insertion/implantation of the prothesis | Discharge Visit, an average of 24h
  Evaluation of surgeon's satisfaction with the usability of the device during the procedure (current implant procedure), the comfort level for insertion/implantation of the prothesis (5 options: Definitely satisfied, Satisfied, Somewhat satisfied, Somewhat dissatisfied, Definitely dissatisfied)
Performance : number of steps of increase in bra cup size | 3 months, 1 year and 2 years post-procedure
  Overall mean number of steps of increase in bra cup size at 3 months, 1 year and 2 years post-procedure
Performance : change in chest circumference at the level of the breasts | 3 months, 1 year and 2 years post-procedure
  Overall mean change in chest circumference at the level of the breasts following the implant procedure analyzed as change in thoracic measure at 3 months, 1 years and 2 years post-procedure
Performance : satisfaction with the implant size choice | 3 months, 1 year and 2 years post-procedure
  Suitability of the implant size choice at the time of the procedure analyzed as the difference between the final decision of the cup size for surgery and the cup size at 3 months, 1 year and 2 years
Performance : global satisfaction of the patient | 3 months, 1 year and 2 years post-procedure
  Evaluation of global patient satisfaction at 3 months, 1 year and 2 years post-procedure with the BREAST EVALUATION QUESTIONNAIRE (BEQ55) (5 options: 1 = Very dissatisfied, 2 = Somewhat dissatisfied, 3 = Neither satisfied nor dissatisfied, 4 = Somewhat satisfied, 5 = Very satisfied)
Performance : global satisfaction of the surgeon | 3 months, 1 year and 2 years post-procedure
  Surgeon satisfaction at 3 months, 1 year and 2 years post-procedure evaluated as :
  * degree of symmetry (4 options: NA, Good, Mediocre, Bad),
  * degree of ptosis (3 options: Good, Mediocre, Bad),
  * quality of contours (3 options: Good, Mediocre, Bad),
  * implant placement (2 options: correct placement, visible deformation of the gel),
  * global satisfaction (5 scoring options : definitely satisfied, satisfied, somewhat satisfied, somewhat dissatisfied and definitely dissatisfied).

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Clinique Urbain V Elsan, Avignon
  - Clinique Saint George, Nice
  - Clinique Sainte Geneviève, Paris
  - Clinique Bizet, Paris
  - Clinique du Rond Point des Champs Elysées, Paris
  - Clinique Charcot, Sainte-Foy-lès-Lyon

IPD SHARING:
Plan to Share IPD: No